CLINICAL TRIAL: NCT06287736
Title: A Novel Neuromodulation Approach to Target Small Fiber Neuropathy Early in Diabetes and Measure Functional Recovery
Brief Title: Spinal Cord Stimulation and Small Fiber Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Neuright, Inc. (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Dalm, Assistant Professor, Neurological Surgery, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023H0386; 1R01DK138849-01 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-03-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Conventional Medical Management (CMM). Group1 (No Intervention)
- Spinal Cord Stimulator (SCS) immediate activation. Group 2 (Active Comparator)
  Interventions: Device: Spinal Cord Stimulator Implantation (SCS)
- Spinal Cord Stimulator (SCS) Delayed activation. Group 3 (Active Comparator)
  Interventions: Device: Spinal Cord Stimulator Implantation (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulator Implantation (SCS) — Spinal cord stimulator implantation is broken up into two parts. The first part involves placement of temporary SCS leads for a one-week trial. If the participants respond favorably to the SCS, then they will undergo the second part and the device is implanted
  Arms: Spinal Cord Stimulator (SCS) Delayed activation. Group 3; Spinal Cord Stimulator (SCS) immediate activation. Group 2

SUMMARY:
This is a prospective randomized control trial. Participants enrolled into the study will be randomized into one of three groups, two of which are treatment groups and the third is a control group. A time course of measurements before and after spinal cord stimulation (SCS) treatment (where applicable) will assess pain, DPN severity, small fiber nerve activity, and metabolic health markers.

DETAILED DESCRIPTION:
Peripheral neuropathy (PN) is caused by diabetes, aging, chemotherapy, and over 30 other conditions, and impacts more than 30 million patients in the US alone. Diabetes is the number one cause of peripheral neuropathy, and more than half of patients with diabetes will eventually develop diabetic peripheral neuropathy (DPN), a complex set of symptoms including pain, numbness, tingling, and burning. Spinal cord stimulation (SCS) is an approved intervention for the treatment of chronic pain, including DPN. Spinal cord stimulation has had FDA approval for the treatment of painful DPN since 2015. This study is being done to learn more about the diagnosis of DPN and treatment of DPN with SCS.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Diagnosis of diabetic peripheral neuropathy refractory to treatment with gabapentin or pregabalin and at least 1 other class of analgesic
* Diagnosis of medically refractory pain secondary to diabetic neuropathy
* Presence of pain for 12 months
* Lower limb pain intensity score ≥4 on a visual analog scale
* DN4 ≥4
* Pass pre-operative neuropsychological assessment (surgical group only)
* Capable of providing informed consent

Exclusion Criteria:

* Severe medical comorbidities that, in the opinion of the surgeon, exclude the patient from surgical intervention
* Spinal disease with severe spinal stenosis or spinal cord compression in the region of the proposed spinal cord stimulator lead placement
* Coagulopathy that cannot be corrected
* Unable to discontinue blood thinning medications
* Hemoglobin A1c level greater than 10
* Presence of systemic infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain level | 18 months post baseline
  change in Visual analog pain scale (VAS). The VAS endpoints range from 'no pain at all' to 'pain as bad as it could be'
Change in Diabetic Peripheral Neuropathy (DPN) Pain using the Neuropathic pain diagnostic questionnaire (DN4) | 18 months post baseline
  Neuropathic Pain Diagnostic "Douleur Neuropathique 4" questionnaire (DN4) is a screening questionnaire to help identify neuropathic pain (NP) in clinical practice and research. It is a clinican-administered questionnaire consisting of 10 items.The first 7 symptoms items are scored by interviewing the patient, and the 3 remaining items are scored by means of clinical examination. The scores are added and a score of 4 or more out of 10 is suggestive of neuropathic pain
Change in PROMIS quality of life in relation to pain level | 18 months post baseline
  Change in patient-reported outcomes measurement (PROMIS 29)

SECONDARY OUTCOMES:
change in neuropathic symptoms using Michigan Neuropathy Screening instrument | 18 months post baseline
  change in Michigan Neuropathy Screening instrument (MNSI). The MNSI is designed to be used in the outpatient setting. The MNSI is broken up into 2 parts. The first part consists of 15 yes/no questions on foot sensation. The highest score is 13, and the higher the score indicates more neuropathic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Dalm, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States